CLINICAL TRIAL: NCT04611607
Title: Cangrelor in Patients With Acute Myocardial Infarction Undergoing PCI After CPR, Ventilated or Cardiogenic Shock
Acronym: CAN-SHOCK
Status: Completed | Type: Observational
Sponsor: IHF GmbH - Institut für Herzinfarktforschung (Other)
Collaborators: Ferrer Internacional S.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: CAN-SHOCK
Record Dates: First submitted 2020-10-15; First posted 2020-11-02 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-03

CONDITIONS: Acute Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This registry will provide information about the efficacy and safety of cangrelor in a very high-risk group of patients with acute myocardial infarction undergoing PCI. It will not only include patients with cardiogenic shock, but a variety of patients not able to swallow tablets, such as those after CPR and/or with invasive or non-invasive ventilation. Therefore it will provide information about the use of cangrelor beyond the current knowledge.

DETAILED DESCRIPTION:
This registry is a non-interventional, multicentre, retrospective cohort study in patients with acute myocardial infarction undergoing PCI after CRP, ventilated and/or with cardiogenic shock.

The study is purely observational; data will be documented retrospectively based on available medical records. No additional data will be collected, no study-related treatment will be initiated.

About 10 - 20 high-volume PCI clinics in Germany treating patients with myocardial infarction are eligible for participation. Participating sites will be given a maximum of 6 months for retrospectively documenting eligible patients.

Eligible are all patients with acute myocardial infarction (STEMI, NSTEMI) who underwent PCI after CRP, ventilated and/or with cardiogenic shock and were treated with cangrelor during index procedure. It is planned to enrol about 400 patients in total. Patient characteristics, procedural details and clinical events occurring during the period between index MI and discharge or death (whichever came first) will be documented based on the relevant existing medical charts of the patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Acute Myocardial infarction (NSTEMI or STEMI)
* PCI with stent implantation
* Treatment with cangrelor during index procedure
* At least one of the following criteria:
* CPR prior to PCI
* Cardiogenic shock
* Heart failure with the need for mechanical or non-invasive ventila-tion

Exclusion Criteria:

No explicit medical exclusion criteria are stated to avoid selection bias.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute myocardial infarction (STEMI, NSTEMI) undergoing PCI and treated with cangrelor after CPR / in cardiogenic shock / with mechanical or non-invasive ventilation
Sampling Method: Non-Probability Sample
Enrollment: 303 (Actual)
Dates: Start 2021-05-04 (Actual); Primary Completion 2022-06-07 (Actual); Study Completion 2022-06-07 (Actual)

PRIMARY OUTCOMES:
Definite stent thrombosis | from procedure for index MI up to 48 hours
  Rate of stent thromboses
Recurrent myocardial infarction | from procedure for index MI up to 48 hours
  Rate of recurrent myocardial infarction according to the universal definition of MI

SECONDARY OUTCOMES:
Definite stent thrombosis | from procedure for index MI until discharge from hospital or intrahosptal death, whichever came first; up to 30 days
  Rate of stent thromboses
Recurrent myocardial infarction | from procedure for index MI until discharge from hospital or intrahosptal death, whichever came first; up to 30 days
  Rate of recurrent myocardial infarction according to the universal definition of MI
Bleeding complications | from procedure for index MI until discharge from hospital or intrahosptal death, whichever came first; up to 30 days
  Rate of bleeding complication according to BARC definition
Mortality | from procedure for index MI until discharge from hospital; up to 30 days
  Rate of death

CONTACTS AND LOCATIONS:
Overall Officials: Uwe Zeymer, Prof, Principal Investigator — Klinikum Ludwigshafen ; Stiftung IHF Institut für Herzinfarktforschung
Locations (10):
- Austria (2):
  - Universitätsklinikum Graz, Graz
  - Klinik Ottakring, Vienna
- Germany (8):
  - Fürst-Stirum Klinikum Bruchsal, Bruchsal
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Klinikum Leverkusen, Leverkusen
  - Klinikum Ludwigshafen, Ludwigshafen
  - Universitätsklinikum Mannheim, Mannheim
  - Hegau-Bodensee Klinikum Singen, Singen
  - Krankenhaus Maria-Hilf, Stadtlohn
  - Universitätsklinikum Tübingen, Tübingen

IPD SHARING:
Plan to Share IPD: No